CLINICAL TRIAL: NCT01585259
Title: A Multi-center, Randomized, Double-blind, Multi-dose Group, Parallel Group and Placebo Controlled Phase Ib-IIa Clinical Study to Evaluate the Safety and Efficacy of Antiplatelet Thrombolysin for Injection for the Treatment of Patients With Non-ST Segment Elevation Myocardial Infarction (NSTEMI).
Brief Title: Anfibatide Phase Ib-IIa Clinical Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lees_Anfibatide_Phase2
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2021-07-14 (Actual); Status verified 2015-07

CONDITIONS: Non-ST Segment Elevation Myocardial Infarction
Keywords: anti-platelet;; safety;; efficacy
MeSH Terms: interventions — agkisacucetin protein, Agkistrodon acutus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anfibatide (Active Comparator): Bolus injection will be finished in 5 minutes immediately when the guidewire passes through the first stenosed vessel; bolus injection of different doses+0.002IU/kg/h intravenous infusion for 48h
  Interventions: Drug: Anfibatide
- Placebo (Placebo Comparator): Bolus injection will be finished in 5 minutes immediately when the guidewire passes through the first stenosed vessel; bolus injection of different doses+0.002IU/kg/h intravenous infusion for 48h
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anfibatide — Snake venom
  Arms: Anfibatide
Drug: Placebo — Saline
  Arms: Placebo

SUMMARY:
Investigate the safety and efficacy of Anfibatide in non-ST segment myocardial infarction patients

DETAILED DESCRIPTION:
1. This study is a phase Ib-IIa exploratory study to observe the safety of Antiplatelet Thrombolysin for Injection for the treatment of non-ST segment myocardial infarction (NSTEMI) patients and preliminarily evaluate the efficacy of different doses, providing the theoretical basis of the phase II and III clinical study protocol.
2. To investigate the pharmacokinetics of different doses.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years;
2. Laboratory tests show increase of the markers of myocardial damage (CK-MB,CTnI), or reduction after increase, with at least one values exceeding the 99th percentile of the upper limit of the reference value;
3. Ischemia symptoms (ischemic chest pain lasts for over 15 minutes, little release after taking nitroglycerin sublingually) or a new myocardial ischemia on electrocardiogram(ECG), i.e. a new ST-T variation (a new or transient depression of ST segment by over 0.1mV, or T-wave inversion≥0.2mV);
4. Patients receive PCI after coronary angiography;
5. Patients, or their family or guardian give signed informed consent forms.

Exclusion Criteria:

1. Patients with severe unstable hemodynamics who should receive urgent PCI;
2. Patients with untreated hypertension (SBP>180 mmHg or DBP >110mmHg) and hypotension shock (SBP<90mmHg/80mmHg for over 30min);
3. Investigator considers patients need to use GPIIb/IIIa receptor antagonists during the study period;
4. After coronary angiography, the number of stenosed vessels >2；lesions in left main branch, severe calcification and artery graft lesions;
5. Patients with heart function in decompensatory phase (Killip grade 3-4) or cardiac shock;
6. Patients with malignant arrhythmia, e.g. the third-degree atrioventricular block, ventricular tachycardia or fibrillation ventricular;
7. Patients with severe hepatic or renal dysfunction, with serum aspartate transaminase(AST) and alanine transaminase (ALT) exceeding 1.5 times the upper limit of reference values, creatinine clearance <30ml/min or serum creatinine ≥200μmol/L or 2.5mg/dl;
8. Patients who have received PCI in the past six months;
9. Patients who have received coronary artery bypass grafting (CABG) previously;
10. Patients who have received invasive operation in the past 3 months;
11. Patients who have suffered from ischemic stroke or transient ischemic attack (TIA) in the past 6 months, or patients with past history of hemorrhagic stroke;
12. Patients who need a long-term treatment of oral anticoagulants (such as warfarin);
13. Patients with active peptic ulcer, or other diseases of hemorrhagic tendency;
14. Patients with disease of coagulation disorder;
15. Hematology test shows platelet count <100,000mm3,or hemoglobin<100g/L;
16. Women in pregnant or lactation period, or women of child-bearing age do not take efficient contraception measures;
17. Patients with an allergic constitution;
18. Patients who is participating in other clinical trials;
19. Patients who do not give a signed informed consent forms;
20. Patients who are not suitable to enroll in the trial according to the investigator's judgement.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Platelet aggregation | up to 48 hours
  The inhibition of ristocetin-induced platelet aggregation as measured by whole blood impedance aggregometr in vitro.
Bleeding events | Day 0 to day 30
  Bleeding events classified according to the Bleeding Academic Research Consortium (BARC) .

SECONDARY OUTCOMES:
Mortality | 30 days after treatment
  all-cause mortality, relapse of nonfatal myocardial infarction, nonfatal stroke, second target vascular reconstructio.
Safety Endpoints | Day 0 to day 30
  Degree of thrombocytopenia; Moderate (<100,000 platelets/mm3); Severe (<50,000 platelets/mm3); Extremely severe (<20,000 platelets/mm3)
Thrombosis formation | 48 hours after infusion during operation
  Thrombosis formation after stent implantation:
Thrombolysis in myocardial infraction (TIMI) | day 0
  The proportion of TIMI from grade 0 to 3 Pre -and post-PCI was evaluated.
Corrected TIMI frame count（CTFC） | day 0
  The values of CTFC were evaluated and compared between groups.
TIMI myocardial perfusion grade （TMBG） | day 0
  The proportion of TMPG from grade 0 to 3 Pre -and post-PCI was evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First hospiatl, Beijing, China

REFERENCES:
- [Derived] Zheng B, Li J, Jiang J, Xiang D, Chen Y, Yu Z, Zeng H, Ge J, Dai X, Liu J, Li B, Huo Y. Safety and efficacy of a platelet glycoprotein Ib inhibitor for patients with non-ST segment elevation myocardial infarction: A phase Ib/IIa study. Pharmacotherapy. 2021 Oct;41(10):828-836. doi: 10.1002/phar.2620. Epub 2021 Sep 21. PMID 34478577